CLINICAL TRIAL: NCT07073937
Title: Three Year Outcomes of Combined Hydrus Microstent With iTrack Canaloplasty
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Craig Chaya, Assistant Professor (Clinical), University of Utah
Other Study IDs: 186645
Record Dates: First submitted 2025-06-20; First posted 2025-07-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Glaucoma, Open Angle; MIGS; Minimally Invasive Glaucoma Surgery; Canaloplasty; Intraocular Pressure (IOP); Cataract Surgery; Surgical Technique; Minimally Invasive Surgical Technique; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Glaucoma patients: Patients from the Moran Eye Center who have open-angle glaucoma and have had a combination of Hydrus and 360-degree canaloplasty with concomitant cataract surgery, who have at least three years of follow-up data.
  Interventions: Other: Retrospective chart review

INTERVENTIONS:
Other: Retrospective chart review — Retrospective study; a total of approximately 100 subjects have been identified to have had minimum 36 months follow-up.

SUMMARY:
The goal of this study is to learn if combining minimally invasive glaucoma surgery (MIGS) procedures with different mechanisms of action increases the effectiveness of MIGS. The main question the study aims to answer is: Does combining viscodilation (a surgical technique, often used in glaucoma treatment, that involves using a high-viscosity, elastic gel to widen and open the Schlemm's canal, a main drainage channel in the eye) with the iTrack catheter, along with the Hydrus microstent, show better reduction in intraocular pressure than cataract surgery alone? Researchers will retrospectively review charts of patients who have open-angle glaucoma who have undergone combination Hydrus implantation and 360-degree iTrack canaloplasty with concomitant cataract surgery, who have at least 36 months of clinical follow-up data. Baseline demographic information and severity of glaucoma will be recorded, as will change from baseline yearly to three years in average optical coherence tomography (OCT) retina nerve fiber layer (RNFL) measurements and visual field (VF) pattern standard deviation. Safety outcomes and the percentage of eyes requiring secondary surgical intervention will be recorded at yearly time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open angle glaucoma (mild, moderate or severe as defined below) who have undergone combined Hydrus and 360 degree canaloplasty with concomitant cataract surgery with at least 3-year follow-up data

  * Mild: Definite optic disc, RNFL, or macular imaging abnormalities consistent with glaucoma and a normal visual field as tested with standard automated perimetry (SAP)
  * Moderate: Definite optic disc, RNFL, or macular imaging abnormalities consistent with glaucoma, and visual field abnormalities in one hemifield that are not within 5 degrees of fixation as tested with SAP
  * Severe: Definite optic disc, RNFL, or macular imaging abnormalities consistent with glaucoma, and visual field abnormalities in both hemifields and/or loss within 5 degrees of fixation in at least one hemifield as tested with standard automated perimetry (SAP)
* Patients who have had prior selective laser trabeculoplasty (SLT) are allowed

Exclusion Criteria:

* Prior corneal graft (penetrating Keratoplasty [PKP], deep anterior lamellar keratoplasty [DALK], Descemet's Stripping Automated Endothelial Keratoplasty [DSAEK], Descemet membrane endothelial keratoplasty [DMEK]) & refractive surgery
* Prior retinal surgery
* Prior MIGS or incisional glaucoma surgery
* Angle closure glaucoma and other secondary glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Moran Eye Center who have open angle glaucoma and have had combination Hydrus and 360 degree canaloplasty with concomitant cataract surgery, who have at least three years of follow up data.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of surgical success at three years. | From baseline to three years post-surgery
  Surgical success is defined as a decrease of one or more glaucoma medications from baseline without an increase in medicated intraocular pressure (IOP).

SECONDARY OUTCOMES:
Mean decrease in IOP from baseline at three years | From baseline to three years post-surgery
Mean number of medication reduction from baseline to three years | From baseline to three years post-surgery
  Mean number of medications the patient has been able to stop taking since baseline
Percentage of eyes with greater than twenty percent reduction in IOP from baseline to year three | From baseline to three years post-surgery
Percentage of eyes that are medication free at three years | At three years post-surgery
  Percentage of eyes that do not need any IOP lowering medication at three years
Percentage of eyes with IOP between 14 and 18 mmHg on the same number of medications or fewer at three years post-surgery | At three years post-surgery
Change in average RNFL from baseline yearly to three years | At baseline, one year, two years and three years post-surgery
  Change from baseline yearly to three years in average optical coherence tomography retina nerve fiber layer measurements. OCT RNFL analysis is a non-invasive imaging technique that measures the thickness of the RNFL to help diagnose and monitor glaucoma.
Change in average HVF PSD from baseline yearly to three years | At baseline, one year, two years and three years post-surgery
  Change from baseline yearly to three years in visual field pattern standard deviation. VF PSD is a metric that measures the irregularity of visual field loss.
Percentage of eyes requiring secondary surgical intervention at yearly time points | At one year, two years and three years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Craig Chaya, MD, Principal Investigator — University of Utah John A. Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No